CLINICAL TRIAL: NCT05218616
Title: Single-dose, Open-label, 2 Periods, 2 Sequences, Randomized Crossover Bioequivalence Study of Aviga 50 mg Capsules (JLLC NATIVITA, Belarus) and Sutent 50 mg Capsules (Pfizer Italia S.R.L.) in Healthy Volunteers Under Fasting Conditions
Brief Title: The Bioequivalence Study of Two Sunitinib Products in Capsules 50 mg in Healthy Volunteers Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JLLC NatiVita (Industry)
Collaborators: National Anti Doping Laboratory, Belarus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BE-50-SNB-2020
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Bioequivalence
Keywords: Sunitinib, Bioequivalence, Aviga
MeSH Terms: interventions — Capsules; Sunitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other)
  Interventions: Drug: Aviga, capsules 50 mg / Sutent®, capsules 50 mg
- Sequence RT (Other)
  Interventions: Drug: Sutent®, capsules 50 mg / Aviga, capsules 50 mg

INTERVENTIONS:
Drug: Aviga, capsules 50 mg / Sutent®, capsules 50 mg — Aviga is manufactured by JLLC NATIVITA, Republic of Belarus. Each capsule contains 50 mg of Sunitinib / Sutent® is manufactured by Pfizer Italia S.R.L., Italia. Each capsule contains 50 mg of Sunitinib.
  Other Names: The test product / The reference product
  Arms: Sequence TR
Drug: Sutent®, capsules 50 mg / Aviga, capsules 50 mg — Sutent® is manufactured by Pfizer Italia S.R.L., Italia. Each capsule contains 50 mg of Sunitinib / Aviga is manufactured by JLLC NATIVITA, Republic of Belarus. Each capsule contains 50 mg of Sunitinib
  Other Names: The reference product / The test product
  Arms: Sequence RT

SUMMARY:
The study is designed in accordance with the Eurasian Economic Union (EAEU) regulatory guidelines, with the aim of characterizing the bioavailability of two pharmaceutical products of sunitinib in healthy adult volunteers. Within the clinical portion of the study, each volunteer will receive a single oral dose of the test and the reference product in compliance with the generated randomization code.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged between 18 to 55 years (incl).
2. Body mass index 18.5-30 kg/m² (incl).
3. No signs of acute or chronic disease during the screening.
4. Laboratory blood and urine values are within the normal range or within 10% of the normal range of deviations and are considered by researchers to be clinically insignificant.
5. Non-smokers or ex-smokers (defined as completely quitting smoking for at least three months prior to being included in the test).
6. No known history of alcohol abuse, intake of fewer than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine, or 50 ml of spirits).
7. No known history of drugs abuse at least 6 months prior to being included in the test (benzodiazepines, opioids, cocaine, barbiturates, marijuana, amphetamine).
8. Willingness to comply with the protocol requirements regarding the restriction of the consumption of foods as well as requirements regarding the intake of food, fluids, and physical activity imposed by the study. Xanthine-containing products (coffee, tea (including tutsan tea), chocolate, cola, cacao, energy drinks, etc.) should be excluded from the diet for at least 48 hours before taking the drug. Products containing tobacco, alcohol-containing products and beverages, concentrated fruit and vegetable juices, grapefruit and/or its juice, other citrus fruits and drinks containing quinine, food containing poppy, fatty, spicy and smoked foods should be excluded at least 72 hours before taking the drug. Cruciferous vegetables (broccoli, Brussels sprouts, cauliflower, kohlrabi, as well as white and red cabbage, savoy, and Chinese cabbage) should be excluded at least 7 days before taking the drug.
9. Healthy subject according to medical history, physical examination, and assessment of basic vital signs.
10. No significant abnormalities on 12-lead ECG.
11. No significant abnormalities on the chest X-ray that was performed within 12 months prior to the start of the study.
12. Volunteer's consent to use two medically effective methods of contraception, at least one of which is a barrier method (from the date of screening to the completion of the study and within 10 weeks after the last dose of drugs).
13. The subject's voluntary willingness to provide written informed consent.
14. The ability, at the judgment of the researcher, to follow all the requirements of the protocol.

Exclusion Criteria:

1. Burdened allergic history.
2. Contraindications for use or hypersensitivity to the active substance or excipients that are part of any of the investigational drugs.
3. The medical need in taking CYP3A4 inhibitors (ketoconazole, ritonavir, itraconazole, erythromycin, clarithromycin), CYP3A4 inducers (rifampicin, dexamethasone, phenytoin, carbamazepine, phenobarbital), within 30 days before the start of the study, including injection of a depot or implant of any drug less than 3 months before the start of the study.
4. Use of any over-the-counter or prescription drugs (including vitamins, minerals, herbal drugs, in particular containing tutsan), use of any dietary supplements less than 14 days before the day of taking the study drug, and throughout the study.
5. Any medical or surgical intervention in history that could disrupt the activity of the hematopoietic system, gastrointestinal tract, urinary, and other body systems.
6. History or presence of significant urinary, cardiovascular, pulmonary, neuroendocrine, immunological, neurological, hematological, gastrointestinal, and other body systems, visual organ, or psychiatric disease or disorder.
7. Any hereditary disease.
8. Participation in any clinical studies less than 90 days prior to the beginning of the current clinical study.
9. Oncological disease at present or in history.
10. Any blood/plasma donation and/or bleeding in the amount of 450 ml, as well as if the volunteers were transfused with whole blood or its components less than 60 days before the start of the study.
11. History or presence of clinically significant hemostasiological disorders or bleeding.
12. Acute infections less than 4 weeks before the start of the study, as well as a positive test result for HIV, syphilis, HBV, and HCV.
13. Positive breath test for alcohol and urinalysis for drugs.
14. Swallowing problems in medical history.
15. Use of prohibited foods and drinks.
16. Subjects with abnormal heart rhythm (HR at rest ≥ 100 bpm or ≤ 50 bpm) and BP (systolic BP ≤100 mmHg or diastolic BP ≤60 mmHg or systolic BP ≥140 mm Hg or diastolic BP ≥ 90 mmHg) on the day of the examination or in the history.
17. Difficulty with taking blood for tests.
18. The values of the parameters of the laboratory and instrumental findings are beyond the normal range (over 10% of the normal range of deviations) or are considered by researchers to be clinically significant.
19. Vegetarianism or any other type of diet.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-01-21 (Estimated); Primary Completion 2022-03-03 (Estimated); Study Completion 2022-05-03 (Estimated)

PRIMARY OUTCOMES:
Cmax of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  The maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  The area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
AUC0-∞ of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  The area under the plasma concentration versus time curve from time 0 to to infinite time
Tmax of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  The time to maximum measured plasma concentration
Kel of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  The elimination rate constant
T1/2 of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  Plasma Elimination Half-Life
AUCresid of sunitinib for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 1; 2; 3; 4; 5; 5,5; 6; 6,5; 7; 7,5; 8; 8,5; 9; 9,5; 10; 10,5; 11; 11,5; 12; 13; 14; 16; 24; 36; 48; 72 hours after dosing
  Residual area under the pharmacokinetic curve from the time of the last measured concentration to infinite time
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | Up to 39 days
  An AE is defined as any untoward medical occurrence in a subject administered the test or the reference product and which does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Anti-Doping Laboratory, Lyasny, Minsk Oblast, Belarus